CLINICAL TRIAL: NCT03633435
Title: Feasibility of a Home HD Program Assisted by a Nurse Coming at Home for Arterio-venous Fistula (AVF) Cannulation
Brief Title: Home Hemodialysis Assisted by a Nurse for Arterio-venous Fistula Cannulation
Acronym: DIADIDEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: NxStage Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00992-53
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hemolysis; Cannulation; Arteriovenous Fistula; Nurse's Role
MeSH Terms: conditions — Hemolysis; Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: All incident and prevalent dialysis patients of our unit will get information on that assisted HHD program and will be able to choose this technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- assisted home hemodialysis patients (Experimental): all patients starting assisted home hemodialysis during the study period
  Interventions: Procedure: assisted home hemodialysis patients

INTERVENTIONS:
Procedure: assisted home hemodialysis patients — Arteriovenous fistula cannulation at the patient's home provided by a trained private nurse at each dialysis session with the rope-ladder technique, and connection to the Nxstage System One

SUMMARY:
Home HD (HHD) is associated with better outcome in end-stage renal disease patients compared to in-center HD, in particular in terms of quality of life. However fear of AVF cannulation is a known barrier for patient's choice and adoption of a HHD program. Providing nurse assistance for the cannulation can help developing HHD programs. The aim of this study is to evaluate the feasibility of assisted home hemodialysis, with the intervention of a nurse at home for arterio-venous fistula cannulation.

DETAILED DESCRIPTION:
* Monocentric prospective interventional study.
* Intervention is assisted HHD, defined as: rope-ladder cannulation at the patient's home provided by a trained private nurse at each dialysis session, and connection to the Nxstage System One
* pilot study, with main objective defined as feasibility of the investigator's assisted HHD program. Pilot study usually concerns a small population, allowing us to develop thereafter a bigger study if the results are encouraging.
* primary end-point criteria defined as definitive cessation of HHD with transfer to an other dialysis modality.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be aged more than 18, able to read and write, and have a person with him at home during HD session, according to the french law.

Exclusion criteria:

* medical contra-indication for HHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
failure of assisted- HDD | 12months
  definitive cessation of HHD with transfer to an other dialysis modality.

CONTACTS AND LOCATIONS:
Locations (1):
- caen University hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided